CLINICAL TRIAL: NCT02993198
Title: A Prospective Study of Early Stage Breast Cancer Patients With Abnormal Myocardial Deformation Treated With Anthracycline and/or Trastuzumab and Pertuzumab-based Cancer Therapy
Brief Title: A Prospective Study of Breast Cancer Patients With Abnormal Strain Imaging
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Nausheen Akhter, Assistant Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU00200675
Record Dates: First submitted 2016-12-02; First posted 2016-12-15 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: HER2 Positive Breast Cancer; Cardiovascular Abnormalities
MeSH Terms: conditions — Cardiovascular Abnormalities | interventions — Carvedilol

ARMS (2):
- Prophylactic Carvedilol (Experimental): Carvedilol 3.125 mg by mouth every 12 hours, titrated to a max dose of 25 mg by mouth every 12 hours, depending on blood pressure and heart rate, until completion of study.
  Interventions: Drug: Carvedilol
- No Therapy (No Intervention): Standard of care monitoring without prophylactic treatment.

INTERVENTIONS:
Drug: Carvedilol
  Arms: Prophylactic Carvedilol

SUMMARY:
The Cardio-Oncology program at Northwestern offers care to cancer patients who develop cardiac toxicities from chemotherapy. Breast cancer patients with the tumor marker for HER2 necessitate treatment with anthracycline and/or trastuzumab and pertuzumab-based chemotherapies, which are known to cause cardiac toxicities. Breast cancer patients will undergo a "cardio-oncology echocardiogram" which incorporates advanced left ventricular assessment by utilizing deformation or strain imaging during chemotherapy treatment for surveillance of cardiac toxicities. The aims of this project are:

1. To create a registry of both clinical, and echocardiographic variables, biomarkers, and genetic analysis that will be used to develop a risk model to predict LV dysfunction in early stage breast cancer patients undergoing chemotherapy with anthracycline and/or trastuzumab and pertuzumab-based chemotherapy regimens.
2. To propose a new management algorithm for initiation of prophylactic beta-blocker therapy for early stage breast cancer patients with preclinical cardiac toxicities demonstrated by strain parameters.
3. To determine if initiation of prophylactic beta-blocker therapy in patients with early cardiac toxicity can delay or prevent a drop in LV EF and the development of clinical heart failure.
4. To explore serial measurements of a suite of novel biomarkers during ongoing anticancer treatment that are presumed but not yet proven to be predictive of cardiac dysfunction in women with breast cancer.
5. To identify DNA biomarkers of predilection to cardiotoxicity.
6. To generate hiPSC to validate markers predictive of cardiotoxicity.

DETAILED DESCRIPTION:
150 patients will be prospectively consented/screened. Over the course of the study, 30 patients are expected to develop abnormal strain with a normal EF > 53%. They will be randomized in 1:1 fashion to open label carvedilol vs. no treatment.

All consenting patients will receive a baseline echocardiogram and blood draw for biomarkers and genetic testing. Patients will be followed with echocardiograms at 3 month intervals for 12 months, until completion of trastuzumab/pertuzumab therapy.

Based on echocardiogram findings, patient will fall into four study arms (A, B, C, D). Patients in Arm A (normal EF and normal strain) and Arm D (decrease in EF > 10%, to a value <53%) will receive current standard of care treatment and will be followed in a registry arm. Arms B and C will comprise of 30 patients with normal EF who develop preclinical cardiac dysfunction, as defined as a change in global longitudinal strain of > 15% from baseline strain) or < -15% absolute longitudinal strain will be prospectively assigned 1:1 to receive prophylactic carvedilol (Arm B) vs. no treatment (Arm C). Prophylactic carvedilol will be initiated at the starting dose of 3.125 mg PO BID and titrated based on blood pressure and heart rate.

Patients will be seen every 3 weeks during the titration phase at their chemotherapy appointments. At each visit, vitals and symptoms will be assessed for dizziness and side-effects from carvedilol. If patient complains of dizziness or HR < 50 bpm, or SBP < 100 mmHg, then the dose titration should stop and the dose should be reduced to the dose at the last increased increment. If there is a > 10% decrease in EF to a value < 53% on the next echocardiogram, then standard heart failure therapy will be initiated (beta-blocker and/or ace-inhibitors) and chemotherapy will be held as per standard of care. If patients require other standard of care treatments for heart failure, such as diuretic therapy or aldosterone antagonists, then this will also be initiated. At this point, these patients will be considered to have met the study endpoint. However, if there is an improvement or no change in strain and EF, then patients will continue with cardiac surveillance with an echo at 3 month intervals. Patients who have been assigned to receive prophylactic carvedilol will continue treatment for duration of chemotherapy up to 1 year. Prophylactic carvedilol will be stopped at the completion of study.

A biomarker substudy will be conducted on 100 patients. These patients will have labs drawn every at ten time points, baseline and every 6 weeks for 12 months, and 1 year post-chemotherapy. A separate blood draw for generation of hiPSC and DNA testing would be done for 100 patients. The blood collection will coincide with the patient's chemotherapy infusions with trastuzumab. These biomarkers will allow for further characterization of patients at risk for developing CTRCD.

A "cardio-oncology" echocardiogram will include standard 2D M-mode and Doppler echocardiography, 2D strain imaging, and 3D LV volume. This data will be processed on-line or off-line within 24 hours of completion of the echocardiogram to determine randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age with HER2-overexpressing early stage breast cancer (Stages I - III)
2. Pathology report must include HER2 expression, estrogen and progesterone receptor status
3. Normal LV function (EF > 53%) on baseline echocardiogram
4. NYHA functional class I-II (no symptoms, dyspnea with more than 2 blocks)
5. Scheduled to receive treatment with anthracycline and/or trastuzumab and pertuzumab-based regimens
6. Patients with a history of HTN, hyperlipidemia, diabetes, mild CAD, mild valvular disease are permitted
7. Patients on concomitant cardiac medications other than beta-blockers (BB) or ace-inhibitors (ACE) therapy are permitted. Other non-cardiac medications are not prohibited.
8. Women of childbearing potential and sexually active men and women should use effective contraception.
9. Patients must have a signed informed consent prior to registration

Exclusion Criteria:

1. LV dysfunction (EF < 53%)
2. New York Heart Association (NYHA) functional class III-IV (heart failure symptoms at less than 2 blocks to advanced symptoms at rest)

   a. NYHA Classification: I - No limitations to activity II - Slight limitation to ordinary activity, no symptoms at rest III - Marked limitation to less than ordinary activity, no symptoms at rest IV - Inability to carry out activity without symptoms, symptoms at rest
3. Pre-existing cardiac disease (moderate-severe coronary artery disease, moderate-severe valvular heart disease, constrictive/restrictive cardiomyopathies)
4. Metastatic breast cancer
5. Patients who have ever taken BB/ACE therapy are excluded.
6. 2nd and 3rd degree AV block
7. Sick sinus syndrome
8. Patients with severe bradycardia (< 50 bpm) or severe hypotension (SBP < 85 mmHg)
9. Severe liver dysfunction defined as Child-Turcotte-Pugh class B & C (significant functional compromise - decompensated disease)
10. Moderate-severe Asthma
11. Hypersensitivity to beta-blockers
12. Patients who are pregnant/lactating are not eligible
13. Unwilling to consent/assent to blood donation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-04; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Global Longitudinal Strain | 1 year
  Improvement or stability in strain from baseline (i.e., increase in strain or decrease by no more than 3%).

SECONDARY OUTCOMES:
Number of cancer treatments | 1 year
  Rate of cancer treatments held for decrement in EF > 10% among groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Gong FF, Grunblatt E, Voss WB, Rangarajan V, Raissi S, Chow K, Jafari L, Patel NP, Vaitenas I, Marion M, Ramirez H, Zhao M, Andrei AC, Baldridge AS, Murtagh G, Maganti K, Rigolin VH, Akhter N. A strain-guided trial of cardioprotection in early-stage breast cancer patients on anti-HER2 therapy (PROTECT HER2). Cardiooncology. 2024 Nov 27;10(1):85. doi: 10.1186/s40959-024-00291-5. PMID 39605014